CLINICAL TRIAL: NCT04534465
Title: A Single Center, Open-label, Parallel Arm, Phase 4 Study to Evaluate the Acceptability of a Prototype Flavor System With Ascending Levels of 2,4,6 Grams or Higher of Mannitol for PEG 3350 Laxative in Subjects Suffering With Occasional Constipation.
Brief Title: Study to Gather Information on the Acceptability of a New Flavor System With Increasing Levels of 2, 4, 6 g or Higher of Mannitol for PEG 3350 in Subjects Having Infrequent Bowel Movements.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18160
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols; polyethylene glycol 3350; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dosing arm 1 (Experimental): MiraLAX Sachet (17g) + Flavor blend (2g mannitol total)
  Interventions: Drug: Polyethylene glycol (MiraLAX, BAY81-8430); Drug: Mannitol
- Dosing arm 2 (Experimental): MiraLAX Sachet (17g) + Flavor blend + additional 2g mannitol (4g mannitol total)
  Interventions: Drug: Polyethylene glycol (MiraLAX, BAY81-8430); Drug: Mannitol
- Dosing arm 3 (Experimental): MiraLAX Sachet (17g) + Flavor blend + additional 4g mannitol (6g mannitol total)
  Interventions: Drug: Polyethylene glycol (MiraLAX, BAY81-8430); Drug: Mannitol
- Dosing arm 4 (Experimental): MiraLAX Sachet (17g) + Flavor blend + additional 6g mannitol (8g mannitol total)
  Interventions: Drug: Polyethylene glycol (MiraLAX, BAY81-8430); Drug: Mannitol
- Dosing arm 5 (Experimental): MiraLAX Sachet (17g) + Flavor blend + additional 8g mannitol (10g mannitol total)
  Interventions: Drug: Polyethylene glycol (MiraLAX, BAY81-8430); Drug: Mannitol

INTERVENTIONS:
Drug: Polyethylene glycol (MiraLAX, BAY81-8430) — Oral solution, 17g polyethylene glycol, one time
Drug: Mannitol — Oral, 2g, 4g, 6g, 8g and 10g mannitol, one time

SUMMARY:
Study to gather information on the acceptability of a new flavor system with increasing levels of 2, 4, 6 g or higher of the sugar alcohol Mannitol for Polyethylene glycol (PEG) 3350 a drug stimulating bowel movement to pass stool in subjects having infrequent bowel movements. The taste of the various preparations will be measured by use of a rating scale.

ELIGIBILITY:
Male and female subjects, aged 18 years and older, suffering with occasional constipation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02-13 (Actual); Primary Completion 2013-03-19 (Actual); Study Completion 2013-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Merck Consumer Center, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in US from 13Feb2013 (first patient first visit) to 19Mar2013 (last patient last visit).
Pre-assignment Details: Sixty-two (62) subjects was screened and fifty (50) subjected completed the study.
Period: Overall Study
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Started | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Population: MiraLAX Sachet (17g) + Flavor blend (2g, 4g, 6g, 8g and 10g mannitol total). Baseline data were not collected separately for Arms/Groups.
Arm/Group | All Population
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: Years] | 43.9 [28 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 25
  Asian | 1
  Caucasian | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Opinion of the Products' Flavor
Description: Evaluated by 7-point scales: 1-extremely dislike, 2-moderately dislike, 3-dislike somewhat, 4-neither like nor dislike, 5-like somewhat, 6-moderately like, 7-extremely like
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Dosiing Arm 3: MiraLAX Sachet (17g) + Flavor blend + additional 4g mannitol (6g mannitol total)
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  1- Extremely Dislike | 1 | 0 | 0 | 0 | 0
  2- Moderately Dislike | 0 | 3 | 0 | 0 | 0
  3- Dislike Somewhat | 1 | 1 | 1 | 0 | 0
  4- Neither Like nor Dislike | 4 | 1 | 4 | 0 | 1
  5- Like Somewhat | 3 | 1 | 2 | 4 | 3
  6- Moderately Like | 0 | 3 | 2 | 4 | 2
  7- Extremely Like | 1 | 1 | 1 | 2 | 4

2. Primary Outcome: Number of Participants With the Opinion of the Amount of Flavor in the Products
Description: Evaluated by 7-point scales: -3 -extremely weak, -2 -somewhat weak, -1 -slightly weak, 0 -just the right level of flavor, 1 -slightly intense, 2 -moderately intense, 3 -much too intense
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  -3 - Extremely Weak | 0 | 0 | 1 | 0 | 0
  -2 - Somewhat Weak | 1 | 1 | 2 | 1 | 0
  -1 - Slightly Weak | 4 | 1 | 3 | 2 | 1
  0 - Just the Right Level of Flavor | 5 | 8 | 3 | 7 | 8
  1 - Slightly Intense | 0 | 0 | 1 | 0 | 1
  2 - Moderately Intense | 0 | 0 | 0 | 0 | 0
  3 - Much Too Intense | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With the Opinion of the Products' Sweetness
Description: Evaluated by 7-point scales: -3 -no sweetness needed, -2 -needs to be moderately sweeter, -1 -needs to be a little sweeter, 0 -just the right level of sweetness, 1 -slightly too sweet, 2 -moderately sweet, 3 -much too sweet
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  -3 - No Sweetness Needed | 0 | 0 | 1 | 1 | 1
  -2 - Needs to be Moderately Sweeter | 1 | 1 | 1 | 0 | 0
  -1 - Needs to be a Little Sweeter | 7 | 6 | 6 | 3 | 2
  0 - Just the Right Level of Sweetness | 2 | 3 | 2 | 5 | 7
  1 - Slightly Too Sweet | 0 | 0 | 0 | 1 | 0
  2 - Moderately Sweet | 0 | 0 | 0 | 0 | 0
  3 - Much Too Sweet | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With/Without Cooling Sensation in the Products.
Description: Whether or not subjects felt a cooling sensation (yes/no).
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Yes | 1 | 1 | 3 | 2 | 3
  No | 9 | 9 | 7 | 8 | 7

5. Secondary Outcome: Number of Participants With no Bowel Movement
Description: The number of subjects who did not report any bowel movement was evaluated.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 1 | 2 | 1 | 1 | 1

6. Secondary Outcome: Time to First Bowel Movement (In Hours)
Description: The mean and standard deviation of the time to first bowel movement in hours were evaluated.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 9 | 8 | 9 | 9 | 9
Hours | 6.672 (6.367) | 5.444 (4.095) | 5.117 (6.987) | 2.470 (1.464) | 4.543 (2.718)

7. Secondary Outcome: Number of Participants for Gas Rating
Description: A gas rating score of 0 means that there was no gas experienced, while a score of 1 represents slight gas experienced, 2 represents moderate gas experienced and 3 represents severe gas experienced.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  0 | 0 | 2 | 2 | 0 | 1
  1 | 4 | 5 | 4 | 3 | 2
  2 | 5 | 1 | 1 | 5 | 3
  3 | 1 | 2 | 3 | 2 | 4

8. Secondary Outcome: Number of Participants for Bloating Rating
Description: A score of zero represents no bloating, while a score of 1 represents slight bloating, 2 represents moderate bloating and 3 represents severe bloating.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  0 | 5 | 5 | 1 | 1 | 4
  1 | 2 | 2 | 5 | 4 | 3
  2 | 2 | 3 | 3 | 3 | 3
  3 | 1 | 0 | 1 | 2 | 0

9. Secondary Outcome: Number of Participants for Abdominal Discomfort Rating
Description: A score of 0 represents no abdominal pain, 1 represents slight abdominal pain, 2 represents moderate abdominal pain and 3 represents severe abdominal pain.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10
Participants
  0 | 3 | 5 | 9 | 4 | 6
  1 | 6 | 3 | 1 | 3 | 3
  2 | 0 | 1 | 0 | 3 | 1
  3 | 1 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With no Successful Bowel Movement
Description: The number of subjects who did not report the successful bowel movement was evaluated.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 7 | 6 | 3 | 5 | 6

11. Primary Outcome: Number of Participants With Different Levels of Cooling Sensation of the Products
Description: Evaluated by 4-point scales: 1 -barely perceptible, 2 -slightly noticeable, 3 -moderately noticeable, 4 -extremely noticeable
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 1 | 1 | 3 | 2 | 3
Participants
  1 - Barely Perceptible | 0 | 0 | 0 | 0 | 1
  2 - Slightly Noticeable | 1 | 0 | 1 | 0 | 2
  3 - Moderately Noticeable | 0 | 1 | 2 | 2 | 0
  4 - Extremely Noticeable | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With the Opinion of Aftertaste in the Products.
Description: Whether or not subjects experienced aftertaste (yes/no).
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Yes | 1 | 4 | 6 | 8 | 5
  No | 9 | 6 | 4 | 2 | 5

13. Primary Outcome: Number of Participants With Different Levels of Aftertaste of the Products
Description: Evaluated by 3-point scales: 1 -slightly noticeable, 2 -moderately noticeable, 3 -extremely noticeable
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 1 | 4 | 6 | 8 | 5
Participants
  1 - Slightly Noticeable | 0 | 3 | 4 | 3 | 4
  2 - Moderately Noticeable | 1 | 1 | 1 | 5 | 1
  3 - Extremely Noticeable | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Time to First Successful Bowel Movement (In Hours)
Description: The mean and standard deviation of the time to first successful bowel movement in hours were evaluated.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 3 | 4 | 7 | 5 | 4
Hours | 4.311 (0.826) | 9.967 (8.870) | 8.462 (9.640) | 3.587 (1.759) | 4.683 (3.340)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event
Description: Including serious adverse events and adverse events.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosiing Arm 3 | Dosing Arm 4 | Dosing Arm 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
participants
  Serious Adverse Event | 0 | 0 | 0 | 0 | 0
  Adverse Event | 6 | 3 | 4 | 7 | 6

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Dosing Arm 1 | Dosing Arm 2 | Dosing Arm 3 | Dosing Arm 4 | Dosing Arm 5
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 4/10 | 7/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dosing Arm 1 (N=10) | Dosing Arm 2 (N=10) | Dosing Arm 3 (N=10) | Dosing Arm 4 (N=10) | Dosing Arm 5 (N=10)
Increased Gas (Gastrointestinal disorders) | 3 | 2 | 2 | 6 | 5
Increased Bloating (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 1
Increased Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1
Watery Stool (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days